CLINICAL TRIAL: NCT05334134
Title: Immunological Mechanisms in Multisystem Inflammatory Syndrome in Children
Brief Title: COVID-19: Immunological Mechanisms in Multisystem Inflammatory Syndrome in Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Ulrikka Nygaard, Primary Investigator, Rigshospitalet, Denmark
Other Study IDs: H-20028631_MIS-C_Immunology
Record Dates: First submitted 2022-03-19; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Multisystem Inflammatory Syndrome in Children; COVID-19; SARS-CoV-2 Infection
Keywords: Multisystem Inflammatory Syndrome in Children
MeSH Terms: conditions — pediatric multisystem inflammatory disease, COVID-19 related; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study seeks to explore immunological mechanisms in patients with Multisystem Inflammatory Syndrome in Children (MIS-C) to improve the understanding of this pathogenesis of this disease.

In a cohort of MIS-C patients diagnosed during the Wild type, Alpha, Delta and Omicron waves, research samples will be analyzed for whole-blood RNA expression, proteomics, inflammatory cytokines, cellular immune populations, autoantibodies, as well as host genetic markers.

DETAILED DESCRIPTION:
BACKGROUND Multisystem inflammatory syndrome in children (MIS-C) is a rare severe complication to SARS-CoV-2 infection in children. Thousands of children worldwide have been hospitalized with this new disease. Yet, the immunological mechanisms are sparsely described.

AIM The project seeks to explore immunological mechanisms in patients with MIS-C.

METHOD From a prospective nationwide cohort of patients with MIS-C from Denmark (May 2020-March 2022), research samples will be investigated for whole-blood RNA expression, proteomics, inflammatory cytokines, metabolomics, cellular immune populations, autoantibodies, as well as host genetic markers allowing for detailed mapping this disease. Samples from MIS-C patients will be compared to patients with bacterial and viral disease, and other inflammatory diseases.

TIME FRAME Sample identification: February 1 2022 to April 1, 2022. Sample analysis: April 1, 2022 to December 31, 2022

PERSPECTIVES New molecular-based tools may lead to improved understanding of the pathogenesis of MIS-C. This could form basis for development of novel diagnostic markers, identification of severe phenotype and therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with MIS-C, according to the CDC criteria aged 0-17 years

Exclusion Criteria:

* Patients from whom patient/parent/legal guardian signed consent is not received

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients fulfilling the diagnostic critieria of MIS-C, according to the CDC
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Immunological mechanisms in MIS-C | Day 0-3 and up to during 24 weeks
  Whole-blood RNA expression at admission and change during recovery

CONTACTS AND LOCATIONS:
Overall Officials: Ulrikka Nygaard, MD PhD, Study Chair — Rigshospitalet, Denmark
Locations (1):
- Ulrikka Nygaard, Copenhagen, Denmark